CLINICAL TRIAL: NCT05790928
Title: AONDA Retrospective Study 1
Brief Title: Air Optix Night and Day Aqua (AONDA) Retrospective Study 1
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLD265-P001
Record Dates: First submitted 2023-03-07; First posted 2023-03-30 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Refractive Ametropia; Hyperopia; Myopia
MeSH Terms: conditions — Hyperopia; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- AONDA DW: Lotrafilcon A contact lenses worn in a daily wear (DW) modality (lenses removed nightly for cleaning) for at least 1 year with monthly replacement.
  Interventions: Device: Lotrafilcon A spherical contact lenses
- AONDA CW: Lotrafilcon A contact lenses worn in a continuous wear (CW) modality (lenses worn continuously including overnight) for at least 1 year with monthly replacement.
  Interventions: Device: Lotrafilcon A spherical contact lenses

INTERVENTIONS:
Device: Lotrafilcon A spherical contact lenses — CE-marked silicone hydrogel contact lenses indicated for the optical correction of refractive ametropia (myopia and hyperopia) in persons with minimal astigmatism that does not interfere with visual acuity
  Other Names: AIR OPTIX Night & Day AQUA; AONDA

SUMMARY:
The purpose of this study is to assess long term performance and safety of AONDA in a real world setting when worn as daily wear or continuous wear for vision correction. This study will be used to support AONDA's marketability in Europe and other locations.

DETAILED DESCRIPTION:
In this retrospective observational study, the subject used AONDA for at least approximately 1 year in either a daily wear (DW) or continuous wear (CW) modality with monthly replacement. For the CW cohort only, 3-year data will be collected, if available.

ELIGIBILITY:
Key Inclusion Criteria:

* Normal eyes, as determined or known by the investigator;
* Manifest refraction cylinder less than or equal to 0.75 diopter (D) in each eye at baseline;
* Best Corrected Visual Acuity (BCVA) of 20/25 Snellen or better in each eye at baseline;
* At the time of the 1-year visit, subject was prescribed and wearing AONDA in both eyes in either a DW or CW modality for at least approximately 1 without changing modality;
* Baseline and 1-year visit chart available;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any recurrent history or active anterior segment infection, inflammation, abnormality, or disease contraindicating regular contact lens wear present at baseline;
* The use of systemic or ocular medications contraindicating regular contact lens wear at baseline;
* History of refractive surgery or irregular cornea;
* Slit lamp findings, including signs of pathological dry eye, that would contraindicate regular contact lens wear at baseline;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll charts following a pre-identified process.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-03-25 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Distance visual acuity at Year 1 - DW Cohort | Year 1
  The subject's chart will be reviewed for a distance visual acuity assessment at 1 year after the baseline exam. The 1-year visit will be defined as a visit which occurred 1 year (-2/+4 months) since baseline, during which period the subject was wearing AONDA, and a contact lens examination was performed. Baseline will be defined as the first office visit where the investigator provided an in-person office biomicroscopy exam to the patient, before or during which a contact lens prescription for AONDA was released.
Distance Visual Acuity at Year 1 - CW Cohort | Year 1
  The subject's chart will be reviewed for a distance visual acuity assessment at 1 year after the baseline exam. The 1-year visit will be defined as a visit which occurred 1 year (-2/+4 months) since baseline, during which period the subject was wearing AONDA, and a contact lens examination was performed. Baseline will be defined as the first office visit where the investigator provided an in-person office biomicroscopy exam to the patient, before or during which a contact lens prescription for AONDA was released.
Distance Visual Acuity at Year 3 - CW Cohort | Year 3
  The subject's chart will be reviewed for a distance visual acuity assessment at 3 years after the baseline exam. The 3-year visit will be defined as a visit which occurred 3 years (-2/+8 months) since baseline, during which period the subject was wearing AONDA and a contact lens examination was performed. The 3-year visit will be applicable only if the chart indicates the subject was wearing AONDA since baseline and 1-year.
Incidence of Corneal Infiltrative Events up to Year 1 - DW Cohort | Up to Year 1
  The subject's chart will be reviewed for corneal infiltrative adverse events occurring after the baseline exam. Baseline will be defined as the first office visit where the investigator provided an in-person office biomicroscopy exam to the patient, before or during which a contact lens prescription for AONDA was released.
Incidence of Corneal Infiltrative Events up to Year 1 - CW Cohort | Up to Year 1
  The subject's chart will be reviewed for corneal infiltrative adverse events occurring after the baseline exam. Baseline will be defined as the first office visit where the investigator provided an in-person office biomicroscopy exam to the patient, before or during which a contact lens prescription for AONDA was released.
Incidence of Corneal Infiltrative Events Up to Year 3 - CW Cohort | Up to Year 3
  The subject's chart will be reviewed for corneal infiltrative adverse events occurring after the baseline exam. Baseline will be defined as the first office visit where the investigator provided an in-person office biomicroscopy exam to the patient, before or during which a contact lens prescription for AONDA was released.
Incidence of Microbial Keratitis up to Year 1 - DW Cohort | Up to Year 1
  The subject's chart will be reviewed for incidences of microbial keratitis occurring after the baseline exam. Baseline will be defined as the first office visit where the investigator provided an in-person office biomicroscopy exam to the patient, before or during which a contact lens prescription for AONDA was released.
Incidence of Microbial Keratitis up to Year 1 - CW Cohort | Up to Year 1
  The subject's chart will be reviewed for incidences of microbial keratitis occurring after the baseline exam. Baseline will be defined as the first office visit where the investigator provided an in-person office biomicroscopy exam to the patient, before or during which a contact lens prescription for AONDA was released.
Incidence of Microbial Keratitis up to Year 3 - CW Cohort | Up to Year 3
  The subject's chart will be reviewed for incidences of microbial keratitis occurring after the baseline exam. Baseline will be defined as the first office visit where the investigator provided an in-person office biomicroscopy exam to the patient, before or during which a contact lens prescription for AONDA was released.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CRD, Study Director — Alcon Research, LLC
Locations (4):
- United States (4):
  - Tallahassee Eye Center, Tallahassee, Florida
  - Franklin Park Eye Center PC, Franklin Park, Illinois
  - The Eye Doctors Inc, Eden Prairie, Minnesota
  - Optometry Group, PLLC, Memphis, Tennessee